CLINICAL TRIAL: NCT03406663
Title: A Korean, Single-center, Open-label, Randomized Study of Two Titration Algorithms With Insulin Glargine 300 Units/mL in Patients With Type 2 Diabetes Mellitus
Brief Title: The Korean TITRATION Study: Comparison of the Self-titration Methods for Glargine-300
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Young Min Cho, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-1708-078-878
Record Dates: First submitted 2017-12-18; First posted 2018-01-23 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): In group 1, the dose of Gla-300 will be titrated by the patients by 1 unit per day until achieving a fasting SMPG in the target range of 4.4 to 5.6 mmol/L (INSIGHT algorithm).
  Titration algorithms:
  Patients will be instructed to daily adjust their dose of Gla-300 based on fasting SMPG values. Fasting SMPG will be measured daily by the patient before breakfast and any intake of antihyperglycemic agents.
  Fasting SMPG in the range of
  1. ≥ 5.6 mmol/L, increase 1 unit of Gla-300 dose
  2. > 4.4 and ≤ 5.6 mmol/L, no change
  3. < 4.4 mmol/L, reduce 1 unit of Gla-300 dose
  Interventions: Behavioral: Group 1
- Group 2 (Active Comparator): In group 2, the dose of Gla-300 will be titrated by the patients based on the SMPG values of the last 3 days at least weekly, but no more often than every 3 days to achieve a fasting SMPG in the target range of 4.4 to 5.6 mmol/L (EDITION algorithm).
  Fasting SMPG (median of the last 3 days including current day) in the range of
  1. ≥ 7.8 mmol/L, increase 6 units of Gla-300 dose
  2. > 5.6 and < 7.8 mmol/L, increase 3 units of Gla-300 dose
  3. > 4.4 and ≤ 5.6 mmol/L, no change
  4. ≥ 3.3 and < 4.4 mmol/L, reduce 3 units of Gla-300 dose
  5. < 3.3 mmol/L or occurrence of ≥ 2 symptomatic or 1 severe hypoglycemic episode in the preceding week, reduce 3 units of Gla-300 dose or at the discretion of the investigator
  Interventions: Behavioral: Group 2

INTERVENTIONS:
Behavioral: Group 1 — Patients will be instructed to daily adjust their dose of Gla-300 based on fasting SMPG values. Fasting SMPG will be measured daily by the patient before breakfast and any intake of antihyperglycemic agents.
  Fasting SMPG in the range of
  ≥ 5.6 mmol/L, increase 1 unit of Gla-300 dose, > 4.4 and ≤ 5.6 mmol/L, no change, < 4.4 mmol/L, reduce 1 unit of Gla-300 dose
  Other Names: INSIGHT algorithm
  Arms: Group 1
Behavioral: Group 2 — Fasting SMPG (median of the last 3 days including current day) in the range of
  * 7.8 mmol/L, increase 6 units of Gla-300 dose, > 5.6 and < 7.8 mmol/L, increase 3 units of Gla-300 dose, > 4.4 and ≤ 5.6 mmol/L, no change,
  * 3.3 and < 4.4 mmol/L, reduce 3 units of Gla-300 dose, < 3.3 mmol/L or occurrence of ≥ 2 symptomatic or 1 severe hypoglycemic episode in the preceding week, reduce 3 units of Gla-300 dose or at the discretion of the investigator
  Other Names: EDITION algorithm
  Arms: Group 2

SUMMARY:
The aim of this study is to demonstrate efficacy and safety of self-titration algorithm with Gla-300 using the INSIGHT algorithm (once daily by 1 unit) and the EDITION algorithm (once weekly by 3 units) in Korean patients with T2D.

DETAILED DESCRIPTION:
The primary objective of this study is to obtain efficacy and safety descriptive data on two different titration algorithms: the INSIGHT titration algorithm (self-titration of 1 unit/day) and the EDITION trial algorithm with insulin glargine 300 units/mL (GLA-300) when given as basal insulin in uncontrolled T2DM patients on basal insulin with or without non-insulin anti-hyperglycemic agent (NIAHA) or in insulin naïve patients.

In a Korean, single-center, type 2 diabetes patients with basal insulin therapy will be enrolled. They will be randomly assigned to either titration algorithm for GLA-300. After 12 weeks, the glycemic control, patients' satisfaction to the titration methods and healthcare providers' satisfaction to titration methods will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 19 years
* Treated for T2D for at least 6 months
* Uncontrolled T2D
* Use of SMPG
* HbA1c > 7% and ≤ 10% in patients with a basal insulin (Gla-100, Gla-300, neutral protamine Hagedorn (NPH), and detemir) or HbA1c > 7% and ≤ 11% in insulin naive patients
* Signed informed consent

Exclusion Criteria:

* Type 1 diabetes mellitus
* Pregnancy or lactation
* Night-shift worker
* Unwilling to inject insulin or perform SMPG
* Treated with insulin other than basal insulin within the previous 3 months
* Not on stable dose of basal insulin (±20%) in the last 3 months
* Initiation or change in dose of oral anti-hyperglycemic agents in the last 3 months
* History of alcohol or drug abuse
* Active cancer or other significant comorbidities which the investigator would make the patients unsuitable for participating in the study
* Any clinically significant laboratory finding which the which the investigator would make the patients unsuitable for participating in the study
* Known drug allergy to insulin
* Not signed informed consent
* Incompletion of the study
* Participating in another clinical trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving fasting SMPG ≤ 5.6 mmol/L without hypoglycemia at 12 weeks | up to 12 weeks

SECONDARY OUTCOMES:
Changes in HbA1c (%) | up to 12 weeks
Fasting plasma glucose (mmol/L) | up to 12 weeks
Fasting SMPG (mmol/L) | up to 12 weeks
7-point SMPG (mmol/L) | up to 12 weeks
Proportion of patients at HbA1c ≤ 7% | up to 12 weeks
Change in insulin dose (IU) | up to 12 weeks
Change in body weight (kilogram) | up to 12 weeks
Hypoglycemia (number of patients) | up to 12 weeks
Adverse events | up to 12 weeks
Patient satisfaction to the insulin titration method (evaluated by prespecified questionnaire: DTSQs) | up to 12 weeks
Health care professionals' satisfaction to the insulin titration methods (evaluated by prespecirfied questionnaire: health care provider treatment satisfaction questionnaire) | up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Young Min Cho, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Bae JH, Ahn CH, Yang YS, Moon SJ, Kwak SH, Jung HS, Park KS, Cho YM. Efficacy and Safety of Self-Titration Algorithms of Insulin Glargine 300 units/mL in Individuals with Uncontrolled Type 2 Diabetes Mellitus (The Korean TITRATION Study): A Randomized Controlled Trial. Diabetes Metab J. 2022 Jan;46(1):71-80. doi: 10.4093/dmj.2020.0274. Epub 2021 Jun 16. PMID 34130445